CLINICAL TRIAL: NCT03001453
Title: Post-surgical Pain Care Pathways During Enhanced Recovery Surgery Using Exparel (Bupivacaine Liposome Injectable Suspension) Plus Bupivacaine With Epinephrine Versus Bupivacaine.
Brief Title: Intraoperative Liposomal Bupivacaine vs. Bupivacaine for Total Hip Replacement Pain Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Hip Institute (Other)
Responsible Party: Principal Investigator, Benjamin Domb, Medical Director, American Hip Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHI-001
Record Dates: First submitted 2016-11-08; First posted 2016-12-23 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Pain, Postoperative
Keywords: Exparel; total hip replacement; bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal bupivacaine (Active Comparator): Periarticular infiltration cocktail of 20cc of liposomal bupivacaine with 20cc of normal saline and 40cc of 0.25% bupivacaine with epinephrine
  Interventions: Drug: Liposomal Bupivacaine; Drug: 0.25% Bupivacaine with epinephrine; Drug: Saline
- Bupivacaine with epinephrine (Active Comparator): Periarticular infiltration cocktail of 60cc of 0.25% bupivacaine with epinephrine
  Interventions: Drug: 0.25% Bupivacaine with epinephrine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 266mg liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: 0.25% Bupivacaine with epinephrine — 0.25% bupivacaine with epinephrine
  Other Names: Marcaine
Drug: Saline — Normal saline
  Other Names: Saline solution
  Arms: Liposomal bupivacaine

SUMMARY:
The purpose of this study is to compare two medications currently injected intra-operatively to help decrease pain after surgery in patients undergoing a primary total hip replacement (THR). The two medications are Exparel® (bupivacaine liposome injectable suspension) plus bupivacaine with epinephrine versus bupivacaine with epinephrine. This study is looking to see if one medication works better than the other in managing post-operative pain after THR. The study hypothesis is that Exparel® plus bupivacaine with epinephrine will demonstrate better pain management in THR patients post-operatively. Both medications are FDA-approved for post-operative analgesia.

DETAILED DESCRIPTION:
All surgeries were performed by the same orthopaedic surgeon. Two groups, one receiving Exparel® (bupivacaine liposome injectable suspension) plus bupivacaine with epinephrine (LB group) and the other receiving bupivacaine with epinephrine (Control group), will be compared using post-operative pain scores, hospital length of stay, time to ambulation, falls, narcotic use, and narcotic-related adverse effects. Aside from hospital length of stay, all outcomes were recorded for up to 72 hours following surgery. An a priori power analysis was performed to calculate the total number of patients that needed to be enrolled to achieve a minimum 90% power, with the threshold of statistical significance set to 0.05. Based on a previous study reporting a mean oral opioid consumption of 57.04mg ± 25.6 at 24 hours post THR, a mean difference of 17.14mg was considered to be clinically significant. Thus, at least 26 patients were necessary in each group for an adequately powered assessment. The diagnosis for osteoarthritis was determined by patient history, physical examination, and imaging findings. Each patient received a thorough explanation of the protocol, and willing patients signed an informed consent form. All patients underwent a personal preoperative education program regarding pre, intra-, and post-procedural information including physical therapy, expectations, discharge goals, home therapy, and pain management. After written consent was collected, the form was sent to the hospital pharmacy for randomization. Envelopes were randomized, sealed, numbered, and given to the pharmacy staff, ultimately dispensing the envelopes to the nurse in the operating room in numerical order. The pharmacy documented the required information, selected medication, and drug accountability forms according to the contents of the envelopes.

A nurse delivered study drugs to the operating room in a sealed, non-descriptive envelope. During the standard anterior approach procedure, an anesthesiologist administered fentanyl or hydromorphone as needed for analgesia. The local anesthetics were administered after reduction of the implants. Patients in the LB group received 20cc liposomal bupivacaine, 40cc 0.25% bupivacaine with epinephrine, and 20cc of normal saline. Each patient in the control group received 60cc of 0.25% bupivacaine with epinephrine. Using a 20-gauge spinal needle, the local anesthetics were injected using a deep tissue administration technique. Structures innervated by the femoral nerve, superior gluteal nerve, or lateral femoral cutaneous nerve were considered suitable for injection. Throughout administration, frequent aspirations were performed to check for blood and minimize the risk of intravascular injection. The patients, surgical team, and floor staff was blinded to the local anesthetic drugs given.

During hospitalization, patients were observed, evaluated and treated according to postoperative protocols. Patients received opioids for pain management as needed, which was routinely documented by hospital staff. Opioids included fentanyl, hydromorphone, oxycodone, codeine, tramadol, morphine, and hydrocodone. All opioid dosages were converted into morphine equivalent dosages for analysis. Each patient began physical therapy within the first 24 hours postoperatively. Patients were discharged when they were able to begin self-care, their pain was controlled utilizing an oral regimen, and they were able to tolerate oral medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo primary unilateral total hip replacement
* Patients diagnosed with hip osteoarthritis
* Patients failed to improve with conservative measures
* Patients willing and able to sign informed consent

Exclusion Criteria:

* Revision total hip replacement
* Bilateral total hip replacement
* Birmingham hip resurfacing
* Patients with hepatic/kidney disease
* Patients with a known allergy to bupivacaine or other local anesthetics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G Domb, MD, Principal Investigator — American Hip Institute
Locations (2):
- United States (2):
  - Adventist Hinsdale Hospital, Hinsdale, Illinois
  - American Hip Institute, Westmont, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perets I, Walsh JP, Mu BH, Yuen LC, Ashberg L, Battaglia MR, Domb BG. Intraoperative Infiltration of Liposomal Bupivacaine vs Bupivacaine Hydrochloride for Pain Management in Primary Total Hip Arthroplasty: A Prospective Randomized Trial. J Arthroplasty. 2018 Feb;33(2):441-446. doi: 10.1016/j.arth.2017.09.013. Epub 2017 Sep 20. PMID 29033152

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Started | 50 | 57
Completed | 50 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine | Total
Number analyzed (Participants) | 50 | 57 | 107
Age, Continuous [Mean (Full Range); unit: years] | 61.9 [41.8 to 80] | 62.4 [33.7 to 82.1] | 62.1 [33.7 to 82.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 21 | 31 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 29.2 [18.6 to 46] | 31 [19.5 to 55.4] | 30.1 [18.6 to 55.4]
Laterality [Number; unit: hips]
  Left | 19 | 30 | 49
  Right | 31 | 27 | 58
Robotic assistance [Count of Participants; unit: Participants] | 42 | 44 | 86
Preoperative opioid prescription [Count of Participants; unit: Participants]
  Codeine | 1 | 0 | 1
  Hydrocodone | 5 | 7 | 12
  Hydromorphine | 0 | 1 | 1
  Oxycodone | 1 | 2 | 3
American Society of Anesthesiologists Grade [Count of Participants; unit: Participants] — Patients were graded based on the American Society of Anesthesiologists Physical Status Classification System. 1 indicates a normal healthy patient, 2 is a patient with a mild systemic disease, 3 is a patient with a severe systemic disease, and 4 is a patient with a severe systemic disease that is a constant threat to life. Grade 1 is considered to be a better outcome while Grade 4 is considered to be a worse outcome.
  Participants
    1 | 8 | 4 | 12
    2 | 26 | 31 | 57
    3 | 16 | 21 | 37
    4 | 0 | 1 | 1
Exercise regularly [Count of Participants; unit: Participants] | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Morphine Equivalent Consumption
Description: All opioid doses were administered to the patient at 12-hour intervals post-surgery. Doses were recorded till either of the following criteria was met, the patient was discharged or the 72-hour post-surgery timeframe ended. The doses were then collected and converted to OMEs, in milligrams.
Time Frame: 72 hours postoperation, divided into six 12-hour periods
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Number analyzed (Participants) | 50 | 57
mg
  0-12 | 35.1 (24.4) | 50.5 (34.5)
  12-24 | 28.0 (17.4) | 29.6 (20.9)
  24-36 | 16.8 (14.9) | 21.0 (20.2)
  36-48 | 20.6 (17.0) | 27.4 (21.2)
  48-60 | 23.7 (19.5) | 15.4 (19.0)
  60-72 | 20.9 (19.6) | 20.7 (13.4)
  Total | 100.3 (74.3) | 121.2 (87.9)

2. Primary Outcome: Change in Patient-reported Visual Analog Scale (VAS) Pain Intensity Score
Description: Patient-reported VAS pain intensity score (0 = no pain, 10 = worst pain possible) will be collected. Mean VAS scores for the 72-hour period were calculated using the cohort's reported average pain scores at each 12-hour interval.
Time Frame: 72 hours post-operation, divided into six 12-hour periods
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Number analyzed (Participants) | 50 | 57
units on a scale | 3.8 (1.6) | 3.7 (1.7)

3. Primary Outcome: Time to Ambulation More Than 20 Feet (in Hours)
Description: The length of time (in hours) until the patient first ambulates more than 20 feet from the time of surgery will be recorded.
Time Frame: from time of surgery until patient first ambulates more than 20 feet or 72 hours post-surgery or patient discharge, whichever comes first
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Number analyzed (Participants) | 50 | 57
hours | 10.9 (8.8) | 14.0 (11.9)

4. Primary Outcome: Length of Stay (LOS, in Days)
Time Frame: From time of surgery until patient is discharged, an average of 1.5 days.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Number analyzed (Participants) | 50 | 57
Hours | 46.0 (26.2) | 44.4 (27.1)

5. Primary Outcome: Number of Patients That Experienced a Fall
Time Frame: 72 hours postoperation
Measure: Number; unit: participants
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Number analyzed (Participants) | 50 | 57
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Bupivacaine With Epinephrine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/57
Other Adverse Events (participants affected / at risk) | 14/50 | 11/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine (N=50) | Bupivacaine With Epinephrine (N=57)
Constipation (General disorders) | 4 | 1
Nausea (General disorders) | 8 | 6
Vomiting (General disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No